CLINICAL TRIAL: NCT04575415
Title: Bevacizumab Plus EGFR Tyrosine Kinase Inhibitors in Chinese Patients With Stage IIIB-IV EGFR-mutant Non-small Cell Lung Cancer: a Prospective,Multicenter, Non-interventional,Real-world Study
Brief Title: Bevacizumab Plus EGFR-TKIs in Chinese Patients With EGFR-mutant NSCLC: a Real-world Study
Acronym: BELLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1905
Record Dates: First submitted 2020-09-08; First posted 2020-10-05 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: NSCLC
MeSH Terms: interventions — Bevacizumab; Erlotinib Hydrochloride; Gefitinib; icotinib; Afatinib; dacomitinib; osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1:Bevacizumab plus Erlotinib/Gefitinib/Icotinib: Patients with EGFR-mutant NSCLC would receive bevacizumab plus first-generation EGFR-TKIs in clinical routine care. Bevacizumab 15 mg/kg or clinical routine dose would be intravenous infusion on day 1 once every 3 weeks. Erlotinib 150 mg tablets once daily or Gefitinib 250mg once daily or Icotinib 125mg three times a day would be administered.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Gefitinib; Drug: Icotinib
- Arm 2:Bevacizumab plus Afatinib/Dacomitinib: Patients with EGFR-mutant NSCLC would receive bevacizumab plus second-generation EGFR-TKIs in clinical routine care. Bevacizumab 15 mg/kg or clinical routine dose would be intravenous infusion on day 1 once every 3 weeks.Afatinib 40 mg or clinical routine dose once daily or Dacomitinib 45mg or clinical routine dose once daily or clinical routine dose would be administered.
  Interventions: Drug: Bevacizumab; Drug: Afatinib; Drug: Dacomitinib
- Arm 3:Bevacizumab plus Osimertinib: Patients with EGFR-mutant NSCLC would receive bevacizumab plus third-generation EGFR-TKIs in clinical routine care. Bevacizumab 15 mg/kg or clinical routine dose would be intravenous infusion on day 1 once every 3 weeks. Osimertinib 80 mg tablets once daily would be administered.
  Interventions: Drug: Bevacizumab; Drug: Osimertinib

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 15mg/kg or clinical routine dose by intravenous drip infusion on day 1 of a 21-day cycle
  Other Names: Avastin
Drug: Erlotinib — Erlotinib 150mg, orally once a day
  Other Names: Tarceva
  Groups: Arm 1:Bevacizumab plus Erlotinib/Gefitinib/Icotinib
Drug: Gefitinib — Gefitinib 250mg, orally once a day
  Other Names: Iressa
  Groups: Arm 1:Bevacizumab plus Erlotinib/Gefitinib/Icotinib
Drug: Icotinib — Icotinib 125mg three times a day
  Other Names: Conmana
  Groups: Arm 1:Bevacizumab plus Erlotinib/Gefitinib/Icotinib
Drug: Afatinib — Afatinib 40 mg or clinical routine dose once daily
  Other Names: Gilotrif
  Groups: Arm 2:Bevacizumab plus Afatinib/Dacomitinib
Drug: Dacomitinib — Dacomitinib 45mg or clinical routine dose once daily
  Other Names: Vizimpro
  Groups: Arm 2:Bevacizumab plus Afatinib/Dacomitinib
Drug: Osimertinib — Osimertinib 80 mg once daily
  Other Names: Tagrisso
  Groups: Arm 3:Bevacizumab plus Osimertinib

SUMMARY:
This study is a prospective, multicenter, real-world study to investigate the efficacy and safety of bevacizumab plus epidermal growth factor (EGFR) Tyrosine Kinase Inhibitors in Chinese Patients With Stage IIIB/IV EGFR-mutant Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:

  1. Signed Informed Consent Form.
  2. Age≥18 years.
  3. Histologically or cytologically documented inoperable, locally advanced (Stage IIIB, IIIC), metastatic (Stage IV) or recurrent non-squamous NSCLC.
  4. An exon 19 deletion mutation or exon 21 L858R mutation in EGFR has been found clinically, with or without EGFR T790M mutation
  5. Eastern Cooperative Oncology Group performance status 0-2 or KPS ≥60
  6. Previous EGFR-TKIs or anti-angiogenic agents or systemic cytotoxic chemotherapy for locally advanced, metastatic or recurrent disease has not been performed.

     Exclusion Criteria:
* Patients who meet any of the following criteria will be excluded from study entry:

  1. Squamous carcinoma or mixed non-small cell lung cancer with squamous component.
  2. Potential hazard for receiving EGFR-TKIs or bevacizumab by clinical evaluations
  3. Previous history of receiving EGFR-TKIs or bevacizumab treatment prior to study enrollment
  4. Suspected or diagnosed leptomeningeal metastases
  5. Chest radiotherapy within 3 months prior to study enrollment
  6. Open surgery within 4 weeks prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically documented inoperable, locally advanced (Stage IIIB, IIIC) or metastatic (Stage IV) non-squamous NSCLC with EGFR exon 19 deletion or/and exon 21L858R mutation, with or without EGFR T790M mutation, who meet the inclusion criteria will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) for bevacizumab plus first-generation EGFR-TKIs by investigator using RECIST v1.1 | This is a real-world study. The estimated median PFS for bevacizumab plus first-generation EGFR-TKIs is 18 months according to previous data.
  To evaluate the efficacy of bevacizumab combined with first-generation EGFR-TKIs in patients with EGFR-mutant NSCLC as measured by investigators
Progression-free survival (PFS) for bevacizumab plus second-generation EGFR-TKIs by investigator using RECIST v1.1 | This is a real-world study. The estimated median PFS for bevacizumab plus second-generation EGFR-TKIs is 20 months according to previous data.
  To evaluate the efficacy of bevacizumab combined with second-generation EGFR-TKIs in patients with EGFR-mutant NSCLC as measured by investigators.
Progression-free survival (PFS) for bevacizumab plus third-generation EGFR-TKIs by investigator using RECIST v1.1 | This is a real-world study. The estimated median PFS for bevacizumab plus third-generation EGFR-TKIs is 22 months according to previous data.
  To evaluate the efficacy of bevacizumab combined with third-generation EGFR-TKIs in patients with EGFR-mutant NSCLC as measured by investigators.

SECONDARY OUTCOMES:
Objective response rate (ORR) by investigator using RECIST v1.1 | Baseline overall tumor assessment can be performed up to 28 days after the first-dose of treatment. Post-baseline assessment will be performed every six weeks until 1st disease progression, through study completion, an average of 2 years.
  To evaluate the efficacy of bevacizumab combined with EGFR-TKIs in patients with NSCLC harbouring activating EGFR mutations, with or without EGFR T790M mutation,as measured by investigators assessed objective response rate using RECIST v1.1
Disease control rate (DCR) by investigator using RECIST v1.1 | Baseline overall tumor assessment can be performed up to 28 days after the first-dose of treatment. Post-baseline assessment will be performed every six weeks until 1st disease progression, through study completion, an average of 2 years.
  Disease control rate (DCR) will be analyzed using similar method as objective response rate.
Overall survival | The primary analysis on overall survival is espected to perform on 48 months of follow-up.
  To evaluate the efficacy of bevacizumab combined with EGFR-TKIs in patients with NSCLC harbouring activating EGFR mutations,with or without EGFR T790M mutation,as measured by investigators assessed overall survival.
Incidence of Treatment-Emergent Adverse Events using CTCAE V5.0 | This is a real-world study. Safety of the combination treatment is expected to perform until the study completion, an average of 1.5 years,according to CTCAE V5.0.
  To evaluate the incidence of Treatment-Emergent Adverse Events of bevacizumab combined with EGFR-TKIs in patients with NSCLC harbouring activating EGFR mutations,with or without EGFR T790M mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhou, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China